CLINICAL TRIAL: NCT04740359
Title: The Effect of Functional Trunk Training on Trunk Control and Upper Extremity Functions in Hereditary Ataxia Patients With Autosomal Recessive
Brief Title: Functional Trunk Training in Ataxia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Sedat Yiğit, Res Asst, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/107
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Ataxia, Spinocerebellar; Ataxias, Hereditary
Keywords: ataxia,rehabilitation,trunk,disabilities
MeSH Terms: conditions — Spinocerebellar Ataxias; Spinocerebellar Degenerations; Ataxia

STUDY DESIGN:
Intervention Model Description: Participants were divided in two groups. Two groups will get two different intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Routine training; mat exercises and perturbation training
  Interventions: Other: Routine training
- Study (Experimental): Trunk training; Functional training, mat exercises and perturbation training
  Interventions: Other: Functional training

INTERVENTIONS:
Other: Functional training — The therapy program was planned for 8 weeks and the sessions were performed in 45 minutes (min) for 3 days a week. The functional reach (forward-lateral-cross), trunk rotation exercises were performed in the sitting positions.(25min) Facilitation of trunk extension and elongation in the prone position (10 min). Thoracic mobilization on exercise ball (10min).
  Arms: Study
Other: Routine training — The therapy program was planned for 8 weeks and the sessions were performed in 45 minutes (min) for 3 days a week. The strengthening exercises were applied on the mat (3x10 for the first 4 weeks and 3x15 repetition for the last 4 weeks). Eyes open-closed perturbation training was performed for trunk control in sitting and standing positions (10 min.).
  Arms: Control

SUMMARY:
The study is to examine the effect of functional trunk training on trunk control and upper extremity functions in patients with autosomal recessive ataxia.

DETAILED DESCRIPTION:
Hereditary ataxias are a group of genetic diseases characterized by slow progressive gait disturbance. In addition, coordination disorders can be seen in extremities, speech and eye movements. Atrophy is common in the cerebellum. Friedreich's ataxia, ataxia telangiectasia, ataxia with vitamin E deficiency, infantile-onset spinocerebellar atrophy and Marinesco-Sjögren syndrome are autosomal recessive hereditary ataxias. The constant main sign of autosomal recessive ataxia is progressive ataxia.

The trunk has an important role on dynamic stabilization for postural reactions and limb movements. A good trunk support enables movements in other parts of the body to occur more regularly. Trunk stabilization is important to support upper and lower extremity movements, to meet the loads, and to protect the spinal cord. The relationship between upper extremity function, daily living activities and trunk functions has been emphasized in many studies but comparative studies about the rehabilitation were very less.

This study is to evaluate the effect o functional trunk training in patients with autosomal recessive ataxia.

ELIGIBILITY:
Inclusion Criteria:

* Without any communication impairment (seeing, hearing, hearing),
* Have not had surgery for the upper and lower extremities in the last 6 months,
* Between the ages of 5 and 18,
* The mental level determined by the pediatrician is sufficient,

Exclusion Criteria:

* Patients who want to leave the study at any stage of the study
* Patients who do not attend regular training

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
The Functional Independence | through of te study, average 8 weeks
  The Functional Independence Scale for Children (WeeFIM) was used determine to independence level.
Trunk impairment | through of te study, average 8 weeks
  The Trunk Disorder Scale (TIS) was used to assess static and dynamic sitting balance and trunk coordination
The severity of ataxia | through of te study, average 8 weeks
  The International Ataxia Rating Scale (ICARS) was used to determine the severity
The quality of life | through of te study, average 8 weeks
  The Children's Quality of Life Scale (PedsQL) was used determine to quality of life level.

SECONDARY OUTCOMES:
Upper extremity functional performance | through of te study, average 8 weeks
  The 9-Hole Peg test was used to evaluate upper extremity performance
Functional Reach Test | through of te study, average 8 weeks
  Functional Reach Test was used determine to dynamic trunk balance

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan kalyoncu üniversitesi, Gaziantep, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freund JE, Stetts DM. Use of trunk stabilization and locomotor training in an adult with cerebellar ataxia: a single system design. Physiother Theory Pract. 2010 Oct;26(7):447-58. doi: 10.3109/09593980903532234. PMID 20649489
- [Background] Van de Warrenburg BP, Bakker M, Kremer BP, Bloem BR, Allum JH. Trunk sway in patients with spinocerebellar ataxia. Mov Disord. 2005 Aug;20(8):1006-13. doi: 10.1002/mds.20486. PMID 15838852
- [Background] Corben LA, Tai G, Wilson C, Collins V, Churchyard AJ, Delatycki MB. A comparison of three measures of upper limb function in Friedreich ataxia. J Neurol. 2010 Apr;257(4):518-23. doi: 10.1007/s00415-009-5352-7. Epub 2009 Oct 13. PMID 19823893
- [Background] Freund JE, Stetts DM, Vallabhajosula S. Relationships between trunk performance, gait and postural control in persons with multiple sclerosis. NeuroRehabilitation. 2016 Jun 30;39(2):305-17. doi: 10.3233/NRE-161362. PMID 27372366